CLINICAL TRIAL: NCT06222320
Title: Can Kinesiotaping Reduce Pain in Rib Fractures?: Randomized Prospective Study
Brief Title: Kinesiotaping Method for Rib Fractures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, İsmail DAL, Assistant Professor Literally: Doctor Teaching Member, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KastamonuU
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Rib Fractures; Pain, Chest
MeSH Terms: conditions — Rib Fractures; Chest Pain | interventions — Athletic Tape; Acetaminophen; dexketoprofen trometamol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping group (Experimental): Kinesiotaping will be applied to patients in this group in addition to painkillers.
  Interventions: Other: Kinesiotaping
- Routine treatment group (Active Comparator): Patients in this group will be administered painkillers routinely in the hospital.
  Interventions: Drug: Painkillers

INTERVENTIONS:
Other: Kinesiotaping — Kinesiotaping will be applied to patients in this group in addition to painkillers. Kinesiotaping is a physical therapy technique used to treat muscle pain. It is performed with kinesiotaping tapes attached to the skin. These bands are removed after 4-5 days.
  Other Names: Kinesio Tape
  Arms: Kinesiotaping group
Drug: Painkillers — Patients in this group will be treated with painkillers consisting of paracetamol and dexketoprofen.
  Other Names: Paracetamol, Dexketoprofen
  Arms: Routine treatment group

SUMMARY:
Kinesiotaping is used as a physiotherapy method to reduce muscle pain. In this technique, kinesiotaping tapes are attached to the relevant parts of the body. Patients experience serious pain in rib fractures. Kinesiotaping technique can potentially reduce pain by contributing to external stabilization of the ribs. In this study, patients with isolated rib fractures will be divided into two groups. The first group will be treated with kinesiotaping technique and routine painkillers. The second group will receive routine painkiller treatment. Pain scores between both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Isolated thoracic injury within the last 24 hours
* Patients aged 18-100 years

Exclusion Criteria:

* Hemothorax and pneumothorax requiring intervention
* Injury severity index>16
* Asthma and COPD
* Tape allergy
* Loss of consciousness (GCS <15)
* Incapacitated patients
* Fracture of rib number 1-3

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Day 4 Visual Analogue Scale Pain Score | 4 days
  Visual analog scale pain score on the 4th day after rib fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Yes
Time Frame: Data will become available persistantly on 1.4.2025.
Access Criteria: Upon reasonable request principal investigator will share the data.

REFERENCES:
- [Derived] Dal I, Bektas O, Kader S, Bodur G. Can Kinesiotaping Reduce Pain in Rib Fractures?: A Randomized Prospective Study. J Pain Res. 2024 Dec 12;17:4239-4247. doi: 10.2147/JPR.S500974. eCollection 2024. PMID 39691747